CLINICAL TRIAL: NCT06603675
Title: Detection and Analysis of Microplastic Subtypes in the Human Respiratory System.
Brief Title: Microplastics in the Human Respiratory System
Status: Not yet recruiting | Type: Observational
Sponsor: Wielkopolskie Centrum Pulmonologii i Torakochirurgii (Other)
Responsible Party: Principal Investigator, Piotr Gabryel, MD, MD, PhD, Wielkopolskie Centrum Pulmonologii i Torakochirurgii
Other Study IDs: MicroLung24; 2023/07/X/NZ7/00906 (Other Grant/Funding Number: Narodowe Centrum Nauki)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Microplastics; Lung Cancer (NSCLC); Lung Transplantation
Keywords: microplastics; lung; respiratory system; lung cancer; transplantation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Lung parenchyma, lymph nodes, and blood samples will be collected from patients undergoing surgery for lung diseases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Environmental pollution from plastics has become a significant global issue, with microplastics-tiny particles resulting from plastic degradation-being increasingly detected in various environments, including aquatic ecosystems, soil, and air. These particles can enter the human body through ingestion or inhalation. Despite growing concerns, little is known about the prevalence and types of microplastics in human lungs. Some studies suggest that microplastics may negatively impact respiratory function and lead to lung diseases. Hypothetically, they could cause inflammation, metabolic disorders, and contribute to lung cancer development. However, research is still in its early stages, and conclusive evidence about the mechanisms linking microplastics to negative health effects is lacking. This study aims to quantify and characterize microplastics in the lung parenchyma and lymph nodes of patients with lung cancer and other respiratory diseases. Tissue samples will be collected during surgeries, and microplastic particles will be detected using FTIR microspectroscopy. The research may contribute to a better understanding of the role of microplastics in the development of respiratory diseases.

DETAILED DESCRIPTION:
Environmental pollution from plastics has become one of the key global challenges, with microplastics-tiny particles resulting from plastic degradation-being increasingly detected in water, soil, and the atmosphere. Microplastics can enter the human body through ingestion or inhalation. According to studies (Prata et al., 2020), there is a risk of microplastics being present in the human respiratory system, raising public health concerns. Although research on microplastics in human lungs is still in its infancy, some preliminary studies suggest a potential link between their presence and decreased respiratory function or lung diseases (Chen et al., 2022). Hypothetically, microplastics could cause inflammatory reactions, disrupt metabolism, and contribute to lung cancer development. Additionally, it is speculated that inhaled microplastics could settle in lung tissue and spread to other organs through lymphatic and blood vessels, but this hypothesis remains unproven.

Given the limited data and the rising prevalence of respiratory disorders, this study aims to quantify and characterize microplastics present in the lung parenchyma and lymph nodes of patients with lung cancer and other respiratory diseases, such as emphysema or interstitial lung diseases. The study also seeks to clarify the role of microplastics in the development of these conditions. In future stages, the research will focus on uncovering the mechanisms through which microplastics affect lung tissues.

The study model involves analyzing lung tissue and lymph node samples from patients undergoing surgeries for lung cancer, emphysema, and interstitial lung diseases. Microplastic particles will be detected using infrared microspectroscopy (μFTIR). Lung parenchyma, lymph nodes, and blood samples will be collected with patient consent during surgery, and tissues will be stored at -80°C for further analysis.

Following established protocols (Jenner et al., 2022), microplastics will be identified using Fourier Transform Infrared (FTIR) spectroscopy. In addition to microplastic analysis, data on patients' medical history, occupational exposure, respiratory function, smoking habits, and COVID-19 history will be collected alongside surgical and histopathological findings.

The study anticipates detecting microplastics in the respiratory tract and identifying their types. It is possible that this research will establish a correlation between the presence of microplastics and the severity of lung diseases, potentially identifying a new risk factor for respiratory illnesses. Future research will delve deeper into the mechanisms through which microplastics may cause harmful health effects.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery for lung cancer, emphysema, interstitial lung diseases, or other respiratory conditions,
* patients undergoing lung transplantation (lungs removed from transplant recipients),
* age 18 years or older,
* ability to provide informed consent.

Exclusion Criteria:

* patients with a history of recent or ongoing chemotherapy, immunotherapy, or radiation therapy,
* inability or unwillingness to provide informed consent,
* previous lung surgeries,
* insufficient tissue or blood samples available for analysis due to technical or procedural reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group comprises patients from the Department of Thoracic Surgery at Poznan University of Medical Sciences, Wielkopolskie Centrum Pulmonologii i Torakochirurgii. Participants include individuals undergoing surgery for lung cancer, other respiratory diseases such as emphysema and interstitial lung diseases, and lung transplantation (lungs removed from transplant recipients). The group includes individuals with diverse backgrounds, varying occupational exposure histories, smoking status (active and passive), e-cigarette use, and different comorbid conditions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of lung microplastics. | Time of surgery (Single time point; microplastic measurement is performed on a lung sample taken during surgery).
  Number of microplastics particles detected per sample of lung tissue or regional lymph nodes obtained from patients during surgery.

SECONDARY OUTCOMES:
Types of lung microplastics. | Time of surgery (Single time point; microplastic measurement is performed on a lung sample taken during surgery).
  Types of microplastics particles detected per sample of lung tissue or regional lymph nodes obtained from patients during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Cezary Piwkowski, MD, Prof., Study Chair — Poznan University of Medical Sciences
Locations (1):
- Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be shared
Time Frame: Beginning 2 months and ending 5 years after the publication of results.
Access Criteria: A proposal that describes planned analyses mjust be submitted to central contact person.

REFERENCES:
- [Background] Zhao J, Zhang H, Shi L, Jia Y, Sheng H. Detection and quantification of microplastics in various types of human tumor tissues. Ecotoxicol Environ Saf. 2024 Sep 15;283:116818. doi: 10.1016/j.ecoenv.2024.116818. Epub 2024 Jul 30. PMID 39083862
- [Background] Field DT, Green JL, Bennett R, Jenner LC, Sadofsky LR, Chapman E, Loubani M, Rotchell JM. Microplastics in the surgical environment. Environ Int. 2022 Dec;170:107630. doi: 10.1016/j.envint.2022.107630. Epub 2022 Nov 13. PMID 36403328
- [Background] Danopoulos E, Jenner LC, Twiddy M, Rotchell JM. Microplastic Contamination of Seafood Intended for Human Consumption: A Systematic Review and Meta-Analysis. Environ Health Perspect. 2020 Dec;128(12):126002. doi: 10.1289/EHP7171. Epub 2020 Dec 23. PMID 33355482
- [Background] Jenner LC, Rotchell JM, Bennett RT, Cowen M, Tentzeris V, Sadofsky LR. Detection of microplastics in human lung tissue using muFTIR spectroscopy. Sci Total Environ. 2022 Jul 20;831:154907. doi: 10.1016/j.scitotenv.2022.154907. Epub 2022 Mar 29. PMID 35364151